CLINICAL TRIAL: NCT06166277
Title: Cardioneuroablation for the Management of Patients With Recurrent Vasovagal Syncope and Symptomatic Bradyarrhythmias: The CNA-FWRD Registry
Brief Title: Cardioneuroablation for Recurrent Vasovagal Syncope and Bradyarrhythmias: The CNA-FWRD Registry
Acronym: CNA-FWRD
Status: Recruiting | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CNA-FWRD
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Vasovagal Syncope; AV Block-2Nd Degree-Type 1; Sinus Pause
Keywords: vasovagal syncope; av block; sinus pause; pacemaker; cardioneuroablation; radiofrequency ablation
MeSH Terms: conditions — Syncope, Vasovagal; Atrial Standstill; Atrioventricular Block

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Awaiting the intervention, medically managed patients will remain in the control group for analysis purposes
- Procedural group: After undergoing successful radiofrequency cardioneuroablation or permanent pacemaker procedures the patient will cross-over to the procedural group for analysis purposes
  Interventions: Procedure: Ablation procedure

INTERVENTIONS:
Procedure: Ablation procedure — Cardioneuroablation procedure or permanent pacemaker placement
  Other Names: Permanent pacemaker placement
  Groups: Procedural group

SUMMARY:
The CNA-FWRD Registry is an international prospective observational multicenter registry of patients with symptomatic vasovagal syncope and bradyarrhythmias managed under routine care by medical therapy and radiofrequency catheter ablation of ganglionated plexi or permanent pacemaker implantation.

DETAILED DESCRIPTION:
The CNA-FWRD Registry is an international prospective observational multicenter registry of patients with symptomatic vasovagal syncope and bradyarrhythmias managed under routine care by medical therapy and radiofrequency catheter ablation of ganglionated plexi or permanent pacemaker implantation. Major inclusion criteria for enrollment are history of VVS or symptomatic bradyarrhythmia, age < 60 years, and evaluation by a physician and discussion about potential candidacy for radiofrequency cardioneuroablation or permanent pacemaker implantation for medically refractory symptoms.

For analysis purposes, patients awaiting the intervention will remain in the "control group" and will cross-over to the "procedural group" after successful completion of radiofrequency cardioneuroablation procedure. The follow-up for the procedure group will start at completion of CNA procedure, but patients who eventually do not get the procedure will stay in the control group until the end of the study, with similar follow-up performed as for the patients undergoing RFCA procedure. If a patient in the control group undergoes permanent pacemaker placement, then the day after the procedure the patient will be removed from the control group for follow up.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic vasovagal syncope or symptomatic bradyarrhythmia refractory to behavioral and medical measures
* age < 60 years

Exclusion Criteria:

* age > 60 years
* intra-/infra-Hisian AV block
* intrinsic sinus node disease
* history of supraventricular tachycardia
* history of ventricular tachycardia
* presence of structural heart disease related
* prior history of catheter ablation
* presence of inheritable arrhythmic conditions
* orthostatic hypotension on HUTT test
* abnormal thyroid function levels
* Proven indication for permanent pacemaker implantation

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with vasovagal syncope or symptomatic bradyarrhythmia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Syncope | 3 years
  Recurrent syncope

SECONDARY OUTCOMES:
Time to first syncopal recurrence | 3 years
  Time to first syncope episode since enrollment
Syncope burden | 3 years
  Number of syncopal episodes
Presyncope burden | 3 years
  Number of pre syncopal episodes
Ablation induced change in heart rate | 1 year
  Delta change in HR between pre-ablation and post-ablation
Complications associated with GP ablation | 1 year
  Major peri-procedural complications
Quality of life before and 12 months after ablation | 1 year
  QoL assessed by survey
Redo-ablation procedures | 3 years
  Redo-ablation procedures for primary outcomes
Atrial arrhythmias | 3 years
  Development of new atrial arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Tolga Aksu, MD, Study Chair — Yepedite University
Locations (1):
- Rush University Medical Centert, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Scanavacca M, Hachul D. Ganglionated Plexi Ablation to Treat Patients with Refractory Neurally Mediated Syncope and Severe Vagal-Induced Bradycardia. Arq Bras Cardiol. 2019 Jul 15;112(6):709-712. doi: 10.5935/abc.20190107. No abstract available. PMID 31314822
- [Result] Aksu T, Gopinathannair R, Bozyel S, Yalin K, Gupta D. Cardioneuroablation for Treatment of Atrioventricular Block. Circ Arrhythm Electrophysiol. 2021 Sep;14(9):e010018. doi: 10.1161/CIRCEP.121.010018. Epub 2021 Sep 1. PMID 34465122
- [Result] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133